CLINICAL TRIAL: NCT00295607
Title: Comparing Efficacy and Safety of Tacrolimus With Steroids or Monoclonal Anti-IL2R Antibody in HCV Positive in Liver Transplantation
Brief Title: Comparing Efficacy and Safety of Tacrolimus With Steroids or Monoclonal Anti-IL2R Antibody in Hepatitis C Virus (HCV) Positive Liver Transplant Patients
Acronym: CHASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FG-506-01-28
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2011-09

CONDITIONS: Hepatitis C; Liver Transplantation
Keywords: Tacrolimus; Liver Transplantation; Immunosuppression; Adult; Treatment Outcome
MeSH Terms: conditions — Hepatitis C | interventions — Tacrolimus; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Tacrolimus; Drug: steroids, monoclonal anti-IL2R antibody
- 2 (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — immunosuppression
  Other Names: Prograf, FK506
Drug: steroids, monoclonal anti-IL2R antibody — immunosuppression
  Arms: 1

SUMMARY:
This is an exploratory study to evaluate the impact of eliminating steroid administration upon viral HCV load at 12 months measured by quantitative serum HCV-RNA determination in patients transplanted for HCV cirrhosis.

DETAILED DESCRIPTION:
A comparison will be made between two regimens which both include tacrolimus, one utilizing standard steroid administration and the second with daclizumab (MAB) avoiding steroids for both prophylactic administration and anti-rejection treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 65 years of age who will undergo primary orthotopic liver or split liver allograft transplantation for HCV-cirrhosis are eligible for the study.
* Patients receiving a cadaveric liver transplant with compatible ABO blood type can be included.

Exclusion Criteria:

* Recipient of multi-organ transplant
* Recipient of an auxiliary graft
* Patient is receiving ABO incompatible graft
* Patients requiring immunosuppressive treatment
* Patients requiring ongoing corticosteroid therapy.
* Patient has significant, uncontrolled concomitant infections and/or severe diarrhoea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer.
* Patient or donor is known to be HIV positive.
* Patient is allergic or intolerant to study medication
* Patient is pregnant or breast-feeding.
* Patient has been previously enrolled in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Viral load of HCV at 12 months post transplantation | 12 months

SECONDARY OUTCOMES:
Biopsy-proven acute rejection | 12 months
Acute rejection | 12 months
Patient and graft survival | 12 months
Incidence of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Physician, Study Director — Astellas Pharma Europe B.V.
Locations (17):
- Prague, Czechia
- France (4):
  - Besançon
  - Lyon
  - Nice
  - Villejuif
- Germany (3):
  - Berlin
  - Hamburg
  - Mainz
- Italy (3):
  - Bologna
  - Genova
  - Modena
- Warsaw, Poland
- Spain (3):
  - Barakaldo
  - Madrid
  - Santiago
- Gothenburg, Sweden
- London, United Kingdom

REFERENCES:
- See also: Link to FDA Website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda